CLINICAL TRIAL: NCT07129148
Title: Study on the Applicability of New Technologies for Diabetes Complication Management Based on Mobile Health and Wearable Devices
Brief Title: Mobile Health and Wearable Devices for Diabetes Complication Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: First Hospital of China Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital of Kunming Medical University (Other); Tianjin Medical University Chu Hsien-I Memorial Hospital (Unknown); Shanghai 6th People's Hospital (Other); Jinjiang Municipal Hospital, Shanghai Sixth People's Hospital Fujian Campus (Unknown); Sinocare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LYEC2024-0331
Record Dates: First submitted 2025-08-06; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus Type 2; Diabetes Mellitus Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control: Traditional Control (Other): Adopt classic doctor-patient interaction management; receive diet and exercise education upon enrollment, self-monitor blood glucose at home and keep a diary.
  Interventions: Other: Device: No specific devices
- Experimental: Wearable Devices + Data Management Platform (Other): On the basis of classic management, wear CGM , load CGM management software, and monitor health data in real time via mobile software.
  Interventions: Other: Device: CGM,CGM management platform
- Experimental:WeChat mini-program Smart Management (Other): On the basis of classic management, use the "Professor Tang" WeChat mini-program for blood glucose recording and diet/exercise management.
  Interventions: Other: Device: "Professor Tang" WeChat Mini-program
- Experimental:Wearable Devices + WeChat mini-program Management (Other): On the basis of classic management, wear CGM or smartbands , and use the "Professor Tang" WeChat mini-program simultaneously for real-time data monitoring and personalized recommendations.
  Interventions: Other: Device: CGM, Smart Bracelet, "Professor Tang" WeChat Mini-program

INTERVENTIONS:
Other: Device: No specific devices — Routine doctor-patient interaction.
  Arms: Control: Traditional Control
Other: Device: CGM,CGM management platform — Wearable monitoring + CGM management platform-assisted administration
  Arms: Experimental: Wearable Devices + Data Management Platform
Other: Device: "Professor Tang" WeChat Mini-program — Mini-program-assisted health management
  Arms: Experimental:WeChat mini-program Smart Management
Other: Device: CGM, Smart Bracelet, "Professor Tang" WeChat Mini-program — Wearable monitoring + mini-program integrated management
  Arms: Experimental:Wearable Devices + WeChat mini-program Management

SUMMARY:
The value of intelligent lifestyle intervention for T2D and its complications has been initially explored, but evidence-based support for the effectiveness of related AI risk prediction models and intervention models remains to be confirmed. The primary objective of this study is to verify the effectiveness of an AI model for predicting the risk of T2D complications based on phenotype, laboratory indicators and wearable device indicators, and to explore the effect and applicability of an intelligent lifestyle intervention model combining wearable devices and smartphones in preventing T2D complications.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Type 2 Diabetes;
2. Aged ≥ 18 years;
3. Able to accept the diabetes management model with AI-assisted management and wearable device monitoring;
4. Able to provide complete lifestyle records, including medical history, medication status, diet, exercise, etc.;
5. Fully understand the purpose, nature, and methods of the study, voluntarily participate in this study, accept a 3-month follow-up, and sign the informed consent form.

Exclusion Criteria:

1. Having severe mental illness or language barriers;
2. Suffering from malignant tumors;
3. Pregnant or lactating women;
4. Suspected active infections (such as active pulmonary tuberculosis, pneumonia, etc.);
5. Severe hepatic and renal insufficiency (alanine transaminase and/or aspartate transaminase > 3 times the upper limit of normal; estimated glomerular filtration rate < 15 mL/min/1.73 m²);
6. A history of definite major adverse cardiovascular events and/or revascularization and/or intravenous thrombolysis and/or endovascular thrombectomy;
7. Uncontrolled hyperthyroidism or hypothyroidism, pituitary-adrenal dysfunction, or other endocrine diseases;
8. Alcoholism or drug addiction;
9. Receiving insulin therapy;
10. Unable to accept new comprehensive intervention technologies for various reasons (such as personal beliefs, economic factors, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline, 1 year
  Between-group differences in HbA1c change (from Central Lab)

CONTACTS AND LOCATIONS:
Locations (1):
- Second Xiangya Hospital of Central South University, Changsha, China

IPD SHARING:
Plan to Share IPD: No